CLINICAL TRIAL: NCT01845272
Title: Open-label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetic Interactions of Candesartan Cilexetil and Amlodipine Besylate in Healthy Male Volunteers.
Brief Title: Pharmacokinetic Interactions of Candesartan Cilexetil and Amlodipine Besylate
Acronym: CCA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_CCA_101
Record Dates: First submitted 2013-04-23; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
MeSH Terms: interventions — candesartan cilexetil; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): single administration : candesartan cilexetil 32mg, qd, 10days(oral).
  combination administration : candesartan cilexetil 32mg and amlodipine 10mg, qd, 10days(oral).
  Interventions: Drug: candesartan cilexetil 32mg, amlodipine 10mg
- Part 2 (Experimental): single administration : amlodipine 10mg, qd, 10days(oral).
  combination administration : candesartan cilexetil 32mg and amlodipine 10mg, qd, 10days(oral).
  Interventions: Drug: candesartan cilexetil 32mg, amlodipine 10mg

INTERVENTIONS:
Drug: candesartan cilexetil 32mg, amlodipine 10mg — Treatment A (candesartan 10 days), at least 4 days wash-out, Treatment B (candesartan + amlodipine 10 days, 2-period, 2-treatment crossover
  Other Names: atacand 32mg, norvasc 10mg
Drug: candesartan cilexetil 32mg, amlodipine 10mg — Treatment A (amlodipine 10 days), at least 4 days wash-out, Treatment B (candesartan + amlodipine 10 days, 2-period, 2-treatment crossover
  Other Names: atacand 32mg, norvasc 10mg

SUMMARY:
This study is designated to evaluate the pharmacokinetic interactions of candesartan cilexetil and amlodipine besylate in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers in the age between 20 and 55 years old(inclusive)
* Body mass index (BMI) in the range of 18.5 to 27 kg/m2(inclusive)
* Available for the entire study period
* Understand the requirements of the study and voluntarily consent to participate in the study

Exclusion Criteria:

* Subjects with a history of gastrointestinal diseases which might significantly change ADME of medicines
* Systolic blood pressure outside the range of 100 to 150 mmHg or diastolic blood pressure outside the range of 60 to 1000 mmHg for male subjects. when screening period
* Subject with symptoms of acute disease within 14days prior to study medication dosing
* Subjects with a history of clinically significant allergies
* Subjects with a hereditary problems, for example, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects whose clinical laboratory test values are outside the accepted normal range(Especially,AST or ALT >1.5 times to normal range or total bilirubin > 1.5times to normal range)
* History of drug abuse
* History of caffeine, alcohol, smoking abuse

  * caffeine(coffee,tea,coke) or grapefruit juice > 4cups/day
  * smoking > 20 cigarettes/day
  * alcohol > 140g/week
* Positive test results for HBs Ab, HCV Ab, Syphilis regain test
* Participation in any clinical investigation within 30days prior to study medication dosing
* Subjects with whole blood donation within 60days, component blood donation within 30days and blood transfusion within 30days prior to study medication dosing
* Subjects considered as unsuitable based on medical judgement by investigators

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of the drug-drug interactions of candesartan and amlodipine | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jae-wook Ko, MD, PhD, Principal Investigator — Samsung Medical Center